CLINICAL TRIAL: NCT04005144
Title: A Phase I Study of Brigatinib With Binimetinib in Advanced ALK- or ROS1-Rearranged Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Brigatinib and Binimetinib in Treating Patients With Stage IIIB-IV ALK or ROS1-Rearranged Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: Takeda (Industry); Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 186517; NCI-2019-02315 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: ALK Gene Rearrangement; Lung Non-Small Cell Carcinoma; Progressive Disease; ROS1 Gene Rearrangement; Stage IIIB Lung Cancer; Stage IIIC Lung Cancer; Stage IV Lung Cancer; Stage IVA Lung Cancer; Stage IVB Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Disease Progression; Lung Neoplasms | interventions — binimetinib; brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (brigatinib, binimetinib) (Experimental): Patients receive brigatinib PO QD and binimetinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Drug: Brigatinib

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK162
Drug: Brigatinib — Given PO
  Other Names: Alunbrig; AP 26113; AP-26113; AP26113

SUMMARY:
This phase I trial studies the side effects and best dose of brigatinib and binimetinib in treating patients with stage IIIB-IV non-small cell lung cancer and a type of gene mutation called a rearrangement in the ALK or ROS1 genes. Brigatinib and binimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of brigatinib in combination with binimetinib in stage IIIB or IV anaplastic lymphoma kinase (ALK) or ROS1 rearranged non-small cell lung cancer (NSCLC) and the recommended phase 2 dose.

SECONDARY OBJECTIVES:

I. To determine preliminary efficacy of brigatinib in combination with binimetinib in any line of treatment.

II. To characterize the pharmacokinetic parameters of brigatinib in combination with binimetinib.

EXPLORATORY OBJECTIVES:

I. To assess circulating tumor deoxyribonucleic acid (DNA) (ctDNA) utility in evaluating treatment response.

II. To evaluate the blockade of downstream signaling indicating response or resistance to treatment of immunohistochemistry (IHC) for phosphatidylinositol 3-kinase (PI3K)/Protein kinase B (AKT)/Mitogen-activated protein kinase (MAPK) pathway activity evaluation.

OUTLINE: This a dose-escalation study.

Patients receive brigatinib orally (PO) once daily (QD) and binimetinib PO twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 6 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytological confirmed stage IIIB/IV NSCLC
* Documented ALK-rearrangement (or ROS1- rearrangement) break-apart fluorescence in situ hybridization (FISH) (in >= 15% or tumor cells), or next generation sequencing assay performed on tumor sample or cell free DNA in a Clinical Laboratory Improvement Act (CLIA)-approved laboratory
* At least one prior ALK or ROS1 targeted tyrosine kinase inhibitor (TKI). With progression or intolerance of most recent regimen
* Dose Escalation Phase Only: At least one prior ALK or ROS1 targeted TKI. With progression or intolerance of most recent regimen.
* Dose Expansion Phase Only: In addition to the criteria in Exclusion Criteria # 3, ALK+ patients with no prior chemotherapy, immunotherapy, radiation therapy or other systemic therapy are also allowed.
* Measurable or evaluable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Age >= 18 years
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Leukocytes >= 3,000/microliter (mcL)
* Absolute neutrophil count >=1,500/mcL
* Platelets >= 75,000/mcL
* Hemoglobin (Hgb) >= 9 gm/dL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) =< 5 x institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 5 x institutional upper limit of normal if there are liver metastases
* Creatinine within normal institutional limits OR
* Creatinine clearance >= 50 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal
* Female participants who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of the study drugs, or
  * Agree to completely abstain from heterosexual intercourse
* Male participants, even if surgically sterilized (i.e., status post-vasectomy), who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of the study drugs, or
  * Agree to completely abstain from heterosexual intercourse
* Negative pregnancy testing required at screening and cycle 1 day 1 for women of childbearing potential
* Ability to understand a written informed consent document, and willingness to sign it
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Participant is deemed by the investigator to have the initiative and means to be compliant with the protocol (treatment and follow-up)

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 7 days for prior TKI and 14 days for chemotherapy or radiation and 30 days for prior immunotherapy before the first dose of treatment
* Prior treatment with either study drug as most recent treatment or prior discontinuation of either study drug due to toxicity
* Known hypersensitivity to any study drug components
* Known history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis
* Known history of myositis
* History of pancreatitis
* History or current evidence of retinal vein occlusion (RVO) or current risk factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes); history of retinal degenerative disease
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

  * Symptomatic chronic heart failure grade >= 2, history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality < 6 months prior to screening except atrial fibrillation and paroxysmal supraventricular tachycardia.
  * Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

    * Myocardial infarction (MI) within 6 months prior to the first dose of brigatinib
    * Unstable angina within 6 months prior to first dose
    * Symptomatic congestive heart failure requiring treatment (New York Heart Association grade >= 2), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality =< 6 months prior to Screening except atrial fibrillation and paroxysmal supraventricular tachycardia
    * Congestive heart failure requiring treatment (New York Heart Association grade >= 2)
    * Left ventricular ejection fraction (LVEF) < 50% as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO)
    * QT interval corrected for heart rate using the Fridericia formula (QTcF) > 480 msec;
    * History of clinically significant atrial arrhythmia
    * Any history of ventricular arrhythmia
    * Cerebrovascular accident or transient ischemic attack within 6 months prior to first dose
* Uncontrolled hypertension defined as persistent elevation of systolic blood pressure >= 150 mmHg or diastolic blood pressure >= 100 mmHg despite current therapy
* History of chronic inflammatory bowel disease or Crohn?s disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) =< 12 months prior to first dose of study treatment
* Impaired gastrointestinal (GI) function or disease that may significantly alter the absorption of binimetinib or brigatinib (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption)
* History of thromboembolic or cerebrovascular events =< 6 months prior to starting study treatment, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis or pulmonary emboli
* Current neuromuscular disorder(s) associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Major surgery =< 3 weeks prior to starting study drugs, or persistent/ongoing side effects of major surgery
* Pregnant or nursing (lactating) women
* Other severe, acute, or chronic medical conditions including uncontrolled diabetes mellitus or psychiatric conditions or laboratory abnormalities that, in the opinion of the investigator, may increase the risk associated with study participation or may interfere with ability to participate actively in the study
* History of another malignancy. Participants with fully resected non-melanoma skin cancer, indolent early stage second malignancies, or who have been disease free for > three years may be eligible following discussion with study principal investigator (PI)
* Any symptomatic brain metastasis

  * Note: Participants previously treated or untreated for this condition who are asymptomatic in the absence of corticosteroid and anti-epileptic therapy are allowed. Brain metastases must be stable for >= 2 weeks, with imaging (e.g., magnetic resonance imaging [MRI] or computed tomography [CT]) demonstrating no current evidence of progressive brain metastases at screening)
* Participants receiving any medications or substances that are inhibitors or inducers of CYP3A enzyme(s) and CYP2C8 within 14 days of enrollment are ineligible
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose | Up to 12 months
  Evaluating the number and frequency of adverse events as determined by the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version (v)5.0 by investigator's assessment will be used to determine the recommended phase 2 dose for future studies.
Number of Participants with Dose Limiting Toxicities | Up to 28 days
  A dose limiting toxicity (DLT) is generally defined as a grade 3 or higher, treatment-related adverse event that is attributable to the study treatment during the first 28 days of therapy (Cycle 1). The dose limiting toxicity will be based on the tolerability observed during cycle 1 of treatment/observation. Adverse events will be assessed by the investigators using NCI-CTCAE v5.0.
Number of Total Treatment-Emergent Adverse Events (AEs) | From treatment initiation through study completion, an average of 1 year
  Treatment Emergent AEs will be defined by the NCI CTCAE v5.0 as AEs newly occuring after the patient has begun study treatment.
Number of Treatment-Emergent Adverse Events by Grade | From treatment initiation through study completion, an average of 1 year
  Severity grade will be defined by the NCI CTCAE v5.0.
Number of Grade 3 or Greater Treatment-Emergent Adverse Events by CTCAE v5.0 | From treatment initiation through study completion, an average of 1 year
  Severity grade will be defined by the NCI CTCAE v5.0.
Number of Serious Treatment-Emergent Adverse Events by CTCAE v5.0 | From treatment initiation through study completion, an average of 1 year
  Severity grade will be defined by the NCI CTCAE v5.0.
Number of Treatment-Emergent Adverse Events with an Outcome of Death by CTCAE v5.0 | From treatment initiation through study completion, an average of 1 year
  Severity grade will be defined by the NCI CTCAE v5.0.
Number of Treatment-Emergent Adverse Events Leading to Discontinuation of Study Treatment | From treatment initiation through study completion, an average of 1 year
  Severity grade will be defined by the NCI CTCAE v5.0.
Number of Treatment-Emergent Adverse Events Resulting in Interruption, Reduction, or Delay of study treatment | From treatment initiation through study completion, an average of 1 year
  Severity grade will be defined by the NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | From treatment initiation through study completion, an average of 1 year
  RECIST v1.1 will be used to determine the overall response rate defined as participants with a complete response (CR) or a partial response (PR). Point estimate and 95% exact binomial confidence interval (CI) will be obtained for ORR.
Median Depth of Response Assessed by RECIST v1.1 | From treatment initiation through study completion, an average of 1 year
  Will be defined as maximal reduction in tumor size based on Response Evaluation Criteria in Solid Tumors (RECIST) measurement. Median and inter-quartile range will be used to describe the depth of response (the maximal reduction in tumor size based on RECIST measurement).
Area Under the Plasma Concentration versus Time Curve (AUC) of Brigatinib | At pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 hours post-dose on days 1 and 15 of cycle 1
  Plasma concentration assessment (pharmacokinetic data) of brigatinib during coadministration with binimetinib will be determined by assay at various timepoints. The assay will be done by Takeda / their designated vendor.
Median Progression Free Survival (PFS) | Up to 6 months
  PFS is measured as the time from start of treatment to time of disease progression at 6 months. Kaplan-Meier method will be used to describe the describe the median PFS with 95% CI.
Median Overall Survival (OS) | Up to 12 months
  Overall Survival is measures as the time from start of treatment to time of death, or lost to follow-up. Kaplan-Meier method will be used to describe the describe the median OS at 12 months with 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Collin Blakely, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No